CLINICAL TRIAL: NCT06916468
Title: Improving Patient Comfort of Vibratory Anesthetic Devices With a Cotton Dampener
Brief Title: Efficacy of Cotton as a Dampener for Vibration Anesthetic Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Bryan Carroll, Physician, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20250017
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-05

CONDITIONS: Patient Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cotton as a dampener for a standard vibratory anesthetic device (Experimental): A standard pen-like Vibratory Anesthetic Device (VAD) with and without cotton will be applied across five anatomical sites (lateral nasal wall, sub-malar region of the cheek, ear helix, lateral neck, and dorsal side of the forearm) of participants. For each anatomical site, one side (either right or left) will receive vibration with cotton, and the opposite side will receive vibration without cotton in a randomized order. The study will be blinded to participants, who will be instructed to close their eyes or look away during the vibration application. After the pairs of VAD applications, patients will report their preference for each treatment condition.
  Interventions: Device: VAD with Cotton Dampener; Device: Vibratory Anesthetic Device (VAD)

INTERVENTIONS:
Device: VAD with Cotton Dampener — A standard pen-like Vibratory Anesthetic Device (VAD) with cotton will be applied across five anatomical sites (lateral nasal wall, sub-malar region of the cheek, ear helix, lateral neck, and dorsal side of the forearm) of participants. For each anatomical site, one side (either right or left) will receive vibration with cotton, and the opposite side will receive vibration without cotton in a randomized order.
Device: Vibratory Anesthetic Device (VAD) — A standard pen-like Vibratory Anesthetic Device (VAD) without cotton will be applied across five anatomical sites (lateral nasal wall, sub-malar region of the cheek, ear helix, lateral neck, and dorsal side of the forearm) of participants.

SUMMARY:
The study aims to determine the effectiveness of cotton as a dampener for vibratory anesthetic devices (VADs) for dermatologic patients. It will compare patient preferences for VAD use with and without cotton across different anatomical sites and identify factors, such as chronic pain or neuropathy status, that may influence these preferences. Finally, the study seeks to generate preliminary data to inform potential modifications to VAD use, optimizing patient comfort in dermatologic procedures

ELIGIBILITY:
Inclusion Criteria:

1. Age range: from 18+
2. Dermatologic patients at Westlake Clinic
3. Consent: Must provide informed consent to participate in the study.
4. Availability: Able to complete the entire study session, which includes testing all sites in a single session

Exclusion Criteria:

1. Broken skin or known peripheral neuropathy on anatomical site of vibration.
2. Allergies: Known allergy or sensitivity to nitrile gloves or cotton

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Carroll, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilkowski CM, Maytin AK, Klatzky RL, Carroll BT. A pilot study comparing the user preference of different forms of mechanical vibration. Arch Dermatol Res. 2024 Jan 10;316(2):69. doi: 10.1007/s00403-023-02797-x. No abstract available. PMID 38197978
- [Background] Sharma P, Czyz CN, Wulc AE. Investigating the efficacy of vibration anesthesia to reduce pain from cosmetic botulinum toxin injections. Aesthet Surg J. 2011 Nov;31(8):966-71. doi: 10.1177/1090820X11422809. Epub 2011 Oct 14. PMID 22001341
- [Background] Gresham KA, Carroll BT. A Simple Elastomer-Pad Vibratory Dampener to Maximize Pain Control of Injections in Patient's Undergoing Dermatological Surgery. Dermatol Surg. 2016 Jun;42(6):788-90. doi: 10.1097/DSS.0000000000000718. No abstract available. PMID 27176866
- [Background] Govas P, Kazi R, Slaugenhaupt RM, Carroll BT. Effect of a Vibratory Anesthetic Device on Pain Anticipation and Subsequent Pain Perception Among Patients Undergoing Cutaneous Cancer Removal Surgery: A Randomized Clinical Trial. JAMA Facial Plast Surg. 2019 Dec 1;21(6):480-486. doi: 10.1001/jamafacial.2019.0733. PMID 31513234

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cotton as a dampener for a standard vibratory anesthetic device
Started | 53
Completed | 53
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cotton as a dampener for a standard vibratory anesthetic device
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.28 (15.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 53
  More than one race | 0
  Unknown or Not Reported | 0
Current Neuropathy [Count of Participants; unit: Participants]
  Yes | 13
  No | 40
Past Neuropathy, Currently Absent [Count of Participants; unit: Participants]
  Yes | 3
  No | 50
Current Chronic Pain [Count of Participants; unit: Participants]
  Yes | 17
  No | 36
Past Chronic Pain, Currently Absent [Count of Participants; unit: Participants]
  Yes | 7
  No | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Preferred the VAD With Cotton as Measured by Patient Report.
Time Frame: Up to 45 mins
Measure: Count of Participants; unit: Participants
Arm/Group | Cotton as a dampener for a standard vibratory anesthetic device
Number analyzed (Participants) | 53
Participants | 47
Statistical Analysis 1: Comparison: Cotton as a dampener for a standard vibratory anesthetic device; Test type: Other; p < 0.001, Binomial test; Comparing preference to 50/50 baseline; Proportion = 86.79

2. Primary Outcome: Number of Participants Who Preferred the VAD Without Cotton as Measured Patient Report.
Time Frame: Up to 45 mins
Measure: Count of Participants; unit: Participants
Arm/Group | Cotton as a dampener for a standard vibratory anesthetic device
Number analyzed (Participants) | 53
Participants | 6
Statistical Analysis 1: Comparison: Cotton as a dampener for a standard vibratory anesthetic device; Test type: Other; p < 0.001, Proportion; Out of the 53 participants , what proportion preferred the device without the cotton dampener on majority of anatomical sites; Proportion = 13.20

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Cotton as a dampener for a standard vibratory anesthetic device
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT06916468/Prot_SAP_000.pdf